CLINICAL TRIAL: NCT02409628
Title: EktoTherix™ Regenerative Tissue Scaffold for Repair of Surgical Excision Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neotherix Limited (Industry)
Collaborators: Lorien Engineering Solutions (a division of GP Strategies Ltd) (Unknown); Smith & Nephew Advanced Wound Management (Unknown); NAMSA (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKT01
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Non-melanoma Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Non-melanoma Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma; Surgical excision; EktoTherix; Secondary intention healing; Acute wound repair; Tissue repair scaffold; Regenerative medicine scaffold; Electrospun scaffold
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EktoTherix (Experimental): One application of the EktoTherix scaffold to a fresh wound resulting from a full thickness excision of skin cancer.
  Interventions: Device: EktoTherix

INTERVENTIONS:
Device: EktoTherix — The EktoTherix scaffold is applied to the fresh wound resulting from a full thickness excision of non-melanoma skin cancer and then bolstered by the application of a non-adhesive foam dressing (discontinued at the first visit); both scaffold and foam dressing are secured in place using a semi-occlusive film dressing. The EktoTherix-treated wound is assessed weekly as per standard of care.

SUMMARY:
The purpose of study is to assess the safety and performance of EktoTherix™ Tissue Repair Scaffold in the treatment of full-thickness, dermatologic wounds created by the surgical removal of non-melanoma skin cancers.

EktoTherix™ is a medical device developed by Neotherix Limited, manufactured by the polymer processing technique of electrospinning. Described as a "tissue scaffold", EktoTherix is placed into the surgical wound to help the patients' own cells repair the wound, enhancing healing and improving quality (including cosmetic outcome). The tissue scaffold is completely absorbed by the body during the healing process, which means that there is no need to remove it when the wound is healed.

All patients recruited into this study are treated with EktoTherix, are seen weekly until they heal and seen again at the final follow-up visit three months post-surgery.

The investigators hypothesise that the use of EktoTherix will increase incidence of complete healing and result in an overall better cosmetic result of the healed wound.

ELIGIBILITY:
Inclusion Criteria:

* Is the patient at least 18 years of age
* Is the patient male, or is not pregnant or lactating and is using contraception
* Has the patient been diagnosed with a non-melanoma skin cancer (basal cell carcinoma BCC or squamous cell carcinoma SCC) for which the chosen therapeutic option is surgical excision followed by secondary intention healing
* Is the excisional wound greater than 10mm x 10mm in size and less than or equal to 35mm x 35mm after any attempt at primary closure
* Does the patient have limited skin laxity which would make primary closure of the surgical excision difficult
* Is the patient able to understand the aims and objectives of the trial and are they willing to consent

Exclusion Criteria:

* Has the patient been diagnosed with any transmittable viral diseases (HIV, Hepatitis B or C)
* Has the patient been diagnosed with, or is it suspected that they have metastatic disease
* Does the patient have a history of malignant melanoma or any concomitant disease likely to impede wound healing
* Has the patient been diagnosed with pre-existing wound infection
* Is the patient taking any medication known to interfere with skin grafts (i.e. warfarin and other anticoagulants, steroids, NSAIDs and immunosuppressants)
* Has the excised wound been entirely treated by primary closure
* Does the patient have a history of any significant cardiac, pulmonary, renal, hepatic, neurological and/ or immune dysfunction that may affect wound healing
* Does the patient know of any allergy to any of the device materials to be used in the trial
* Does the patient have a known history of poor compliance with medical treatment
* Has the patient participated in this trial previously and healed or been withdrawn
* Is the patient currently participating in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Incidence of device related adverse events | 3 months
  The primary endpoint of the study is to demonstrate the safety of the EktoTherix Tissue Repair Scaffold through the incidence of device related adverse events identified during the study, including clinical infection, whether the wound has healed by the final clinical assessment and any clinically significant laboratory results at three month post-surgery assessment.

SECONDARY OUTCOMES:
Cosmesis (cosmetic outcome is assessed by the Vancouver Burn Scar Assessment Scale (VBSAS) score (clinician's assessment) and by a Visual Analogue Scale (VAS) | 3 months
  The cosmetic outcome is assessed by the Vancouver Burn Scar Assessment Scale (VBSAS) score (clinician's assessment) and by a Visual Analogue Scale (VAS) score (patient's assessment). The VBSAS scale assigns a numerical score by summing individual ratings for pigmentation, vascularity, pliability and height or depression of the wound or scar. The VAS score is a number, between the worst (0) and the best (ten) cosmetic outcome, representing the patient's perception of the treatment.
  The cosmetic outcome is evaluated when the wound is healed (if prior to or on Day 42 Post-surgery Assessment) and at the 3 Month Post-surgery Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Calum C Lyon, BSc BA MA MB BChir MRCP FRCP, Principal Investigator — York Teaching Hospital NHS Foundation Trust; Michael J Raxworthy, BSc PhD MBA, Study Director — Neotherix Limited
Locations (3):
- United Kingdom (3):
  - The James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough, North Yorkshire
  - Scarborough Hospital, York Teaching Hospital NHS Foundation Trust, Scarborough, North Yorkshire
  - The York Hospital, York Teaching Hospital NHS Foundation Trust, York, North Yorkshire

REFERENCES:
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734